CLINICAL TRIAL: NCT02732418
Title: A Study to Evaluate Suppression of Ovulation Following a Single Subcutaneous Administration of Various Doses of Depo-Provera CI
Brief Title: Lower Dose Depo Provera® Contraceptive Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 834119
Record Dates: First submitted 2016-03-30; First posted 2016-04-08 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Contraception
Keywords: CI-contraceptive injection; DMPA-Depot medroxyprogesterone acetate; MPA-Medroxyprogesterone Acetate; subQ-subcutaneous
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Depo-Provera CI 45 mg (Experimental): a single subcutaneous (SC) injection of 45 mg/0.3 mL
  Interventions: Drug: Depo-Provera CI
- Depo-Provera CI 75 mg (Experimental): a single subcutaneous (SC) injection of 75 mg/0.5 mL
  Interventions: Drug: Depo-Provera CI
- Depo-Provera CI 105 mg (Experimental): a single subcutaneous (SC) injection of 105 mg/0.7 mL
  Interventions: Drug: Depo-Provera CI
- Depo-subQ 104 (Active Comparator): a single subcutaneous (SC) injection of 104 mg/0.65 mL
  Interventions: Drug: Depo-subQ 104

INTERVENTIONS:
Drug: Depo-Provera CI — The active ingredient in Depo-Provera is Medroxyprogesterone acetate (MPA)
  Other Names: Depo Provera® Contraceptive Injection
  Arms: Depo-Provera CI 105 mg; Depo-Provera CI 45 mg; Depo-Provera CI 75 mg
Drug: Depo-subQ 104 — The active ingredient in Depo-Provera is Medroxyprogesterone acetate (MPA). Depo-subQ provera 104® (medroxyprogesterone acetate injectable suspension, 104 mg/0.65mL) for subcutaneous injection
  Other Names: depo-subQ provera 104®
  Arms: Depo-subQ 104

SUMMARY:
This is a randomized, partially-blinded, multi-center, parallel-group study to evaluate and compare the PD and PK of MPA after a single SC injection of either 45 mg/0.3 mL, 75 mg/0.5 mL or 105 mg/0.7 mL of Depo-Provera CI, and one cycle of Depo-subQ 104 use when injected in the abdomen, in women of reproductive age with confirmed ovulatory baseline cycle

DETAILED DESCRIPTION:
This is a randomized, partially-blinded, multi-center, parallel-group study to evaluate and compare the PD and PK of MPA after a single SC injection of either 45 mg/0.3 mL, 75 mg/0.5 mL or 105 mg/0.7 mL of Depo-Provera CI, and one cycle of Depo-subQ 104 use when injected in the abdomen, in women of reproductive age with confirmed ovulatory baseline cycle. Baseline ovulation will be confirmed in all women by measuring serum progesterone (P) approximately twice a week during the 2-3 weeks preceding expected menses. Between 48 and 60 participants (12-15 per group) with confirmed ovulation who meet other eligibility criteria will be enrolled and randomized to receive a single SC injection in the abdomen of 1 of 3 doses of Depo-Provera CI: 45 mg/0.3 mL, 75 mg/0.5 mL or 105 mg/0.7 mL or a single dose of Depo-subQ Provera (104 mg/0.65mL). Participants will be followed for 32 weeks (7.5 months) after the injection During the study participants will provide blood samples for MPA, P and estradiol (E2) prior to injection and then frequently at predefined time points through 7.5 months. In addition, for more accurate ascertainment of the PD response we will perform transvaginal ultrasound (TVS) and assess cervical mucus at predefined time points through 7.5 months. Information on adverse events and concomitant medications will be collected throughout the study. Information on acceptability will be collected at predefined time points through 7.5 months.

ELIGIBILITY:
Inclusion Criteria:

* has typical menstrual cycle of 24 to 35 days
* has confirmed ovulatory cycle during the pretreatment phase (serum progesterone ≥ 4.7 ng/mL in 2 consecutive samples)
* is sterilized or using non hormonal intrauterine device (IUD)
* is in good general health as determined by a medical history and physical examination
* 18 to 40 years of age (inclusive)
* willing to provide informed consent and follow all study requirements
* has negative urine pregnancy test and has no desire to become pregnant in the subsequent 12 months
* has a body mass index (BMI) of 18.0 to 35.0 kg/m2, inclusive
* has hemoglobin ≥10.5 g/dL

Exclusion Criteria:

* has medical contraindications to depot medroxyprogesterone acetate (DMPA) [16]
* has undiagnosed mass in breast
* used DMPA in the past 12 months
* used a combined injectable contraceptive in the past 6 months
* used any of the following medications within 1 month prior to enrollment:

  * any investigational drug
  * prohibited drugs per protocol
  * oral contraceptives
  * Nuva-ring
  * contraceptive patch
  * levonorgestrel intrauterine system (LNG IUS) or contraceptive implant
* has been pregnant within last 3 months
* Is currently lactating
* in the opinion of the investigator, is potentially at elevated risk of HIV infection (HIV-positive partner, IV drug use by self or by partner)
* has more than one male sexual partner
* is using or plans to use prohibited drugs per protocol in the next 9 months
* has known sensitivity to MPA
* plans to move to another location in the next 9 months
* has any condition (social or medical), which in the opinion of the investigator would make study participation unsafe, would interfere with adherence to the clinical study requirements or complicate data interpretation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Time to ovulation | 32 weeks after receiving drug
  Time to ovulation indicated by time to reach rupture of the lead follicle based on transvaginal ultrasound (TVS) findings followed by serum progesterone level of >=4.7 ng/mL. The primary objective will be assessed by estimating the cumulative probability of return to ovulation through Month 7.5 from start of therapy in each test group based on the Kaplan-Meier product-limit method, with 95% confidence intervals derived using the complementary log-log transformation.

SECONDARY OUTCOMES:
Measurement of serum MPA concentrations | 32 weeks after receiving drug
  Measure of Peak Concentrations (Cmax)
Time to maximum serum concentration of MPA | 32 weeks after receiving drug
  Time to reach peak concentration of MPA(Tmax)
Occurrence of adverse events | 32 weeks after receiving drug

CONTACTS AND LOCATIONS:
Overall Officials: Vera Halpern, MD, Principal Investigator — FHI 360
Locations (3):
- Universidade Estadual de Campinas (UNICAMP), Campinas, Brazil
- Instituto Chileno De Medicina Reproductiva (ICMER), Santiago, Chile
- Asociación Dominicana Pro Bienestar de la Familia, Inc. (PROFAMILIA), Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data